CLINICAL TRIAL: NCT04557761
Title: Comparison of microMend® Devices to Sutures in Closing Lacerations in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital of Orange County (Other)
Collaborators: KitoTech Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1912154
Record Dates: First submitted 2020-09-02; First posted 2020-09-22 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Laceration; Skin Wound; Wound Heal
Keywords: Laceration; Wounds; Wound dehiscence; Wound healing
MeSH Terms: conditions — Lacerations; Wounds and Injuries | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Closure with microMend® Arm (Experimental): The microMend® wound closure product will be used to close the Subject's laceration. The wound will be covered with a non-stick dressing.
  Interventions: Device: microMend®
- Closure with Sutures Arm (Active Comparator): The Subject's laceration will be closed with sutures. The standard method for suture closed wounds will be followed in accordance with regular institutional policies and procedures.
  Interventions: Device: Closure with Sutures

INTERVENTIONS:
Device: microMend® — microMend® is a novel wound closure device that consists of arrays of tiny staples, known as Microstaples, which are attached to a backing material that is the size and shape of a butterfly closure. The Microstaples enable secure attachment of the device to the skin, allowing for the safe closure of wounds associated with surgery and traumatic injuries, such as lacerations. microMend is listed with the FDA and is available for sale in the United States.
  Arms: Closure with microMend® Arm
Device: Closure with Sutures — The Subject's laceration will be closed with sutures per regular institutional policies and procedures.
  Arms: Closure with Sutures Arm

SUMMARY:
This study will gather information on the use of microMend® to repair lacerations in children and compare the efficacy of microMend® to sutures for laceration repair. microMend® has previously been shown to be less painful and easier to use than sutures, which are the current standard of care for primary wound closures. Results of this research will inform how the treatment of laceration repairs in the pediatric patient population.

DETAILED DESCRIPTION:
Lacerations are typically closed with sutures, staples, tissue adhesives, or bandages. These methods come with several limitations, however. Sutures and staples can be painful, cause inflammation that can lead to scarring, and require return clinic visits for their removal. Tissue adhesives cannot be used to close wounds under tension, can be associated with inflammation, and carry a risk of wound dehiscence. Bandages are also only useful for closing superficial wounds under low tension. Therefore, there is a need for improved products to close wounds associated with laceration repair.

The current study will use a prospective randomized controlled design to compare the use of sutures to microMend® to treat lacerations among children 7-17 years. Performance of sutures and microMend® will be assessed by investigators, providers and subjects. Participants will be randomized 1:1 between closure of lacerations with microMend® or sutures. Results from this study will help gather further information on the use of microMend® to close wounds in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing a laceration repair that would require sutures, staples, or tissue adhesives to close the skin wound.
* Age between 7 and 17 years old
* Written informed consent obtained from Subject or Subject's legal representative
* Ability of Subject to comply with the requirements of the study

Exclusion Criteria:

* Wound in extensor or flexor surface of knee or elbow
* Wound on concave areas of the face, such as orbit of the nasal sidewall
* Wound on fingers or toes
* Wound under high tension
* Wound that has a gap of more than 1 cm between the wound edges immediately prior to application of microMend devices
* Facial or body hair that could impede application of the wound closure device
* Wound with significant tissue injury
* Wound with active bleeding
* Wound where adjacent skin is wet
* Visual evidence of active infection, contaminated or devitalized tissue, or rash at laceration location
* Wound that contain a foreign body
* Wound site that contains tattoo or other identifiable features
* Subject with keloid(s)
* Medical disorder that, in the opinion of the Investigator, could have a significant effect on wound healing
* Pregnancy
* Inability of Subject to carry out Subject instructions
* Subject lacks the capacity to consent
* Currently using medication that, in the opinion of the Investigator, could have a significant effect on wound healing
* Skin disorder, such as psoriasis, or current dermatitis or eczema at wound site
* History of keloids or scar hypertrophy
* Known bleeding diathesis
* Sensitivity or allergy to adhesives or medical tape
* Active infection in any part of the body
* Use of sutures or staples to close underlying skin layers
* Use of staples to close skin wound
* Use of tissue adhesive or other adhesives directly over the wound

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Investigator's Assessment of Wound Closure Device (Questionnaire) | During wound-closure performance
  The investigator will complete a questionnaire about the wound. The questionnaire will capture information about the wound including the cause of laceration, approximate length of the wound, and whether subcutaneous sutures were used prior to application of micro Mend or sutures. The questionnaire will also indicate whether local anesthesia was used.
Investigator's Assessment of Wound Closure Device (Survey) | During wound-closure procedure
  The investigator will rate the performance of the wound closure device using a survey to rate the ease of use, speed of use, wound appearance, and provide an overall rating for the experience of using the wound closure device. Each parameter will be determined to be Excellent, Good, Fair or Poor, which correspond to numerical ratings of 4, 3, 2, and 1, respectively.

SECONDARY OUTCOMES:
Total Procedure Time | During wound-closure procedure
  The investigator or designee will record the total procedure time from the initiation of anesthesia (if used) to completion of closure of the laceration.
Wound Closure Time | During wound-closure procedure
  The investigator or designee will record the time of the wound closure portion of the procedure measured from initiation of first suture or microMend application to completion of the closure.
Subject assessment of level of pain during wound closure procedure | The VAS Score for level of pain during the wound closure procedure will be collected on the day of the wound closure procedure (Study Day 0).
  The Visual Analogue Pain Scale (VAS) is used to measure endpoints on a scale of 0 to 10, with 0 and 10 representing both extremes. To perform the evaluation, the Subject is asked to place a mark on a straight line that has a 0 on the left end and a 10 on the right end of the line. A score of 0 will indicate no pain, while a score of 10 indicates the worst pain imaginable.
Comparison of Provider's rating of wound closure results with microMend to suture | 1 month after wound-closure procedure
  The provider will compare wound closure results between microMend and sutures at the first return clinic visit.
Subject assessment of level of stress during wound closure procedure | The VAS Score for level of stress during the wound closure procedure will be collected on the day of the wound closure procedure (Study Day 0).
  The VAS Score is used to measure endpoints on a scale of 0 to 10, with 0 and 10 representing both extremes. To perform the evaluation, the Subject is asked to place a mark on a straight line that has a 0 on the left end and a 10 on the right end of the line. A score of 0 will indicate no stress, while a score of 10 indicates the worst stress imaginable.
The VAS Score for level of stress during the wound closure procedure will be collected on the day of the wound closure procedure (Study Day 0). | The VAS Score for level of pain during removal of the wound closure device will be collected at the First Return Clinic Visit, Day 5 (5-7) for facial lacerations or Day 8 (7-10) for lacerations elsewhere on the body.
  The VAS Score is used to measure endpoints on a scale of 0 to 10, with 0 and 10 representing both extremes. To perform the evaluation, the Subject is asked to place a mark on a straight line that has a 0 on the left end and a 10 on the right end of the line. A score of 0 will indicate no pain, while a score of 10 indicates the worst pain imaginable.
Subject assessment of level of stress during removal of wound closure device | The VAS Score for level of stress during removal of the wound closure device will be collected on the day of the wound closure procedure (Study Day 0).
  The VAS Score is used to measure endpoints on a scale of 0 to 10, with 0 and 10 representing both extremes. To perform the evaluation, the Subject is asked to place a mark on a straight line that has a 0 on the left end and a 10 on the right end of the line. A score of 0 will indicate no stress, while a score of 10 indicates the worst stress imaginable.
Visual Assessment of wound in individual Subjects taken both before and after application of wound closure device | Photographs will be taken both before and after application of the wound closure device on the day of the wound closure procedure (Day 0). Photographs will be reviewed by an Independent Plastic Surgeon to assess wound appearance and cosmetic results.
  At least two (2) photographs of each wound will be taken before and after application of wound closure device. An Independent Plastic Surgeon will rate wound appearance and cosmetic results on a 0-10 scale, where 10 indicates the best possible appearance and results, while a score of 0 indicates the worst possible results.product.
Visual Assessment of wound in individual Subjects taken both before and after removal of wound closure device | Photographs will be taken both before and after removal of the wound closure device on the day of the wound closure procedure (Day 5-7 for facial lacerations, Day 7-10 for lacerations elsewhere on the body). Photographs will be reviewed by an Independent
  At least two (2) photographs of each wound will be taken before and after application of wound closure device. An Independent Plastic Surgeon will rate wound appearance and cosmetic results on a 0-10 scale, where 10 indicates the best possible appearance and results, while a score of 0 indicates the worst possible results.
Visual Assessment of wound after 1 Month | A minimum of two photographs of each wound will be taken 1 month after initial application of the wound closure device. Photographs will be reviewed by an Independent Plastic Surgeon to assess wound appearance and cosmetic results.
  At least two (2) photographs of each wound will be taken 1 month after initial application of the wound closure device. An Independent Plastic Surgeon will rate wound appearance and cosmetic results on a 0-10 scale, where 10 indicates the best possible appearance and results, while a score of 0 indicates the worst possible results.
Visual Assessment of wound after 3 Months | A minimum of two photographs of each wound will be taken 3 months after initial application of the wound closure device. Photographs will be reviewed by an Independent Plastic Surgeon to assess wound appearance and cosmetic results.
  At least two (2) photographs of each wound will be taken 3 months after initial application of the wound closure device. An Independent Plastic Surgeon will rate wound appearance and cosmetic results on a 0-10 scale, where 10 indicates the best possible appearance and results, while a score of 0 indicates the worst possible results.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore W Heyming, MD, Principal Investigator — CHOC Children's Hospital of Orange County
Locations (1):
- CHOC Children's, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No